CLINICAL TRIAL: NCT02052011
Title: Ranolazine and Microvascular Angina by PET in the Emergency Department (RAMP-ED)
Brief Title: Ranolazine and Microvascular Angina by PET in the Emergency Department
Acronym: RAMP-ED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1312013144
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-02

CONDITIONS: Microvascular Angina
Keywords: Chest Pain; Microvascular Angina; Ranolazine; Emergency department; PET
MeSH Terms: conditions — Microvascular Angina; Chest Pain; Emergencies | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Subjects will take extended release Ranolazine for 4 weeks. Subjects will take 500 mg twice daily for the first week and then 1000 mg twice daily for remaining period (Dosing will be adjusted with concomitant use of diltiazem, verapamil, erythromycin, simvastatin or metformin).
  Interventions: Drug: Ranolazine
- Placebo Control (Placebo Comparator): Subjects will take placebo pill twice daily for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Subjects will take the extended-release Ranolazine for a total of 4 weeks. Subjects will take 500 mg twice daily for the first week and then 1000 mg twice daily for remaining period (Dosing will be adjusted with concomitant use of diltiazem, verapamil, erythromycin, simvastatin or metformin).
  Other Names: Ranexa
  Arms: Intervention Group
Drug: Placebo
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to determine the effectiveness of Ranolazine for the treatment chest pain from disease of small vessels of the heart also known as 'microvascular angina'.

DETAILED DESCRIPTION:
The Yale Chest Pain Center (CPC) is a unique clinical lab that provides an integrated interdisciplinary research team, access to high volume of chest pain patients largely free of coronary disease (93%) as well state of the art diagnostics including cardiac PET and a sophisticated system for serum processing and banking facilities. The CPC cohort represents a unique population with unrecognized microvascular disease and is often only accessible through the ED. We propose a one-year pilot study to understand the mechanisms of angina relief by Ranolazine (n=20) in patients with microvessel disease in the ED population as compared to controls (n=10) at baseline and at 1-month. In addition, changes in pain scores and function as measured by Seattle Angina Questionnaire (SAQ), recidivism and costs will be measured and correlated with changes in coronary flow reserve (CFR). Serum samples will be obtained and banked for future marker analysis as intermediate surrogates of outcomes.

Primary aim: To compare changes in coronary flow reserve as measured by cardiac PET in patients receiving Ranolazine versus controls.

Secondary aim: To determine if Ranolazine changes Seattle Angina Questionnaire (SAQ) scores in association with changes in Coronary Flow Reserve (CFR) versus controls.

Exploratory aim: To compare composite rate of return visits (office, emergency department and hospitalization) for chest pain within 4-weeks of enrollment between patients with and without Ranolazine.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Yale ED CPC
* ≥ 30 years age
* chest pain or angina equivalent as their chief complaint within 24 hours of enrollment
* Coronary Flow Reserve(CFR) <2.5 on PET scan in the ED.

Exclusion Criteria:

* Acute coronary syndrome
* Prior evidence of obstructive heart disease (history of Percutaneous Transluminal Coronary Angioplasty (PTCA), Coronary Artery Bypass Grafting (CABG) or calcium score > 10 on PET scan)
* Resting blood pressure of systolic >180/110 mm Hg or <100/40
* known cardiomyopathy or heart failure
* currently on dialysis
* creatinine clearance <30 ml/min
* liver cirrhosis
* significant aortic stenosis (murmur on exam)
* active use of cocaine or amphetamine
* current use of potent CYP3A4 inducers or inhibitors (such as ketoconazole, clarithromycin, HIV protease inhibitors)
* baseline QTc > 580 msec
* use of drugs that prolong QTc (Haldol, erythromycin)
* pregnancy
* inability to read or understand English
* suffering from a condition that precludes interview (i.e. cognitive or communication impairment).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basmah Safdar, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Safdar B, D'Onofrio G, Dziura J, Russell RR, Johnson C, Sinusas AJ. Ranolazine and Microvascular Angina by PET in the Emergency Department: Results From a Pilot Randomized Controlled Trial. Clin Ther. 2017 Jan;39(1):55-63. doi: 10.1016/j.clinthera.2016.12.002. Epub 2017 Jan 9. PMID 28081848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from June, 2014-November, 2015 at the Yale New Haven Hospital Chest Pain Center, an ED observation unit that treats low-moderate cardiac risk patients.
Period: Overall Study
Arm/Group | Intervention Group | Placebo Control
Started | 21 | 10
Completed | 17 | 8
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo Control | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7) | 50 (5) | 50 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 18 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 14 | 8 | 22
  More than one race | NA — not asked | NA — not asked | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | 0
TIMI Score [Count of Participants; unit: Participants] — Thrombolysis in Myocardial Infarction (TIMI) Score measures mortality risk for unstable angina and myocardial infarction. The score ranges 0-7 with lower score indicating lower risk. 0-2 is considered low risk for acute coronary syndrome.
  Participants
    0-1 | 16 | 9 | 25
    2-3 | 5 | 1 | 6
    4-7 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Coronary Flow Reserve
Description: Compare changes in coronary flow reserve as measured by cardiac PET(Positron Emission Tomography) in patients receiving Ranolazine versus control. This is the ratio between stress and rest myocardial blood flow in response to stress.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Intervention Group | Placebo Control
Number analyzed (Participants) | 17 | 8
ratio
  Baseline CFR | 1.6 (0.3) | 1.6 (0.3)
  Post-Treatment CFR | 1.9 (0.4) | 1.6 (0.4)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.08 to 0.62]

ADVERSE EVENTS:
Arm/Group | Intervention Group | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 3/21 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=21) | Placebo Control (N=10)
Dizziness (General disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Small sample size with higher than expected dropout rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No